CLINICAL TRIAL: NCT05519332
Title: Percutaneous Vertebral-disc Plasty for Thoracolumbar Very Severe Osteoporotic Vertebral Compression Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiawei Jiang (Other)
Responsible Party: Sponsor-Investigator, Jiawei Jiang, resident physician, Affiliated 2 Hospital of Nantong University
Organization: Affiliated 2 Hospital of Nantong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JJiang
Record Dates: First submitted 2022-08-24; First posted 2022-08-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Osteoporotic Fracture of Vertebra
Keywords: percutaneous vertebroplasty; percutaneous cement discoplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVDP group (Experimental): Patients underwent percutaneous vertebral-disc plasty
  Interventions: Procedure: percutaneous vertebral-disc plasty
- PVP group (No Intervention): Patients underwent conventional percutaneous vertebroplasty

INTERVENTIONS:
Procedure: percutaneous vertebral-disc plasty — percutaneous vertebroplasty combined percutaneous cement discoplasty
  Arms: PVDP group

SUMMARY:
Purpose: To compare the clinical outcomes and radiological parameters of patients undergoing percutaneous vertebroplasty (PVP) versus those undergoing percutaneous vertebral-disc plasty (PVDP) for back pain, segmental instability, and kyphosis due to thoracolumbar very severe osteoporotic vertebral compression fractures (vsOVCFs).

This prospective study included elderly patients with thoracolumbar vsOVCFs. All the patients were randomly allocated into the PVP group (who underwent conventional PVP) and the PVDP group (who underwent PVP combined percutaneous cement discoplasty). The visual analogue scale (VAS), Oswestry Disability Index (ODI), local kyphosis angle, and disc height were recorded preoperatively and postoperatively.

DETAILED DESCRIPTION:
Patients diagnosed with thoracolumbar vsOVCFs in hospital and undergoing minimally invasive treatment from November 2019 to March 2021 were enrolled for the study. They were randomly allocated into two groups (based on random numbers generated by www. randomizer.org), namely PVP group and PVDP group.

Operative technique：In PVDP group, PVP and PCD both used a unilateral transpedicular approach into the vertebrae and disc. . Under general anesthesia, the patient was turned over to a prone position, and the deformity is reduced with a slight closed manipulative. Firstly, under fluoroscopic O-arm guidance, the puncture site was localized into the junction made by the transverse process and the superior articular process and entered the target area according to the puncture angle and depth measured before the operation. Secondly, the other puncture cannula was inserted into the intervertebral disc space adjacent to the ruptured endplate through the transpedicular access, and the target area was the middle of the intervertebral space. Thin-cut CT images were obtained intraoperatively by the O-arm fluoroscopy to confirm puncture needle placement location. Third, the bone cement was injected into the vertebrae and the intervertebral disc space, meanwhile, the cannula was also needed to move back to the vertebrae, and the bone cement in the vertebrae could connect the intervertebral disc space and the vertebrae to form a whole. Finally, the PVP group and the adjacent vertebrae performed by prophylactic vertebroplasty used bilateral pedicle puncture, under the guidance of the O-arm, two puncture needles were percutaneously inserted into the vertebrae, reaching about the middle of the vertebrae. Then, cement was slowly injected into the vertebral body, once cement leakage into the spinal canal or veins was detected, the injection was stopped.

The investigators measured radiological parameters including the local kyphotic angle (LKA), disc height anterior (DHA), and disc height posterior (DHP) from lateral plain radiographs preoperatively and at 1 day and final follow-up after surgery. The visual analog score (VAS) was used to assess the preoperative and postoperative back pain relief. The Oswestry Disability Index (ODI) was used to assess the quality of life and was recorded preoperatively, postoperatively, and final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* bone mineral density T scores <-2.5;
* compression of the vertebral anterior column greater than two-thirds of their original height;
* Kyphosis with LKA greater than 20°;
* the accordion phenomenon: the different angles of a supine CT scan and a lateral standing X-ray measurement;
* upper or lower vertebral endplate fracture;
* the involved vertebral body was intact;
* Elderly patients with a history of major illness (such as cardiovascular disease, cancer or active malignancy) and were intolerant of the traditional open surgery.

Exclusion Criteria:

* Pathological vertebral fractures caused by spinal tumors, spinal tuberculosis, and spinal infection and so on;
* Patients with symptoms of nerve roots or spinal cord compression;
* Patients with a previous history of spinal fusion;
* A history of abnormal bleeding or coagulation disorder dysfunction.

Ages: 58 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline visual analogue scale | One day before operation, one day after operation and 1year.
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100. A higher score indicates greater pain intensity. Based on the distribution of pain Visual Analogue Scale scores in post-surgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Visual Analogue Scale have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Change from Baseline Oswestry Disability Index | One day before operation, one day after operation and 1year.
  The ODI assesses ten aspects of daily functions viz. pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. An ODI of 0-20% indicates minimal disability; the patients can cope with most living activities and usually no treatment is indicated, apart from advice on lifting, sitting and exercise. An ODI of 21-40% indicates moderate disability; the patients experience more pain and difficulty with sitting, lifting and standing; travel and social life are more difficult and they may be disabled from work; personal care, sexual activity and sleeping are not grossly affected. An ODI of 41-60% indicates severe disability; pain remains the main problem in this group of patients; the activities of daily living are affected. Patients with an ODI of 61-80% are severely crippled in function with back pain impinging on all aspects of the patient's life. Finally, an ODI of 81-100% indicates that the patients are bed-bound.
Change from Baseline the local kyphotic angle | One day before operation, one day after operation and 1year.
  The local kyphotic angle (LKA) was calculated by a measurement called Cobb's method, which measured the angle between the superior endplate of the upper vertebrae and the inferior endplate of the lower vertebrae. Use this to assess the degree of local kyphosis of the spine.

SECONDARY OUTCOMES:
Change from Baseline the disc height anterior | One day before operation, one day after operation and 1year.
  Disc height anterior(DHA) was measured from the anterior points of the disc on lateral plain radiographs. It is used to assess the degree of height loss at the anterior border of the intervertebral space.
Change from Baseline the disc height posterior | One day before operation, one day after operation and 1year.
  Disc height posterior (DHP) was measured from the posterior points of the disc on lateral plain radiographs. It is used to assess the degree of height loss at the posterior border of the intervertebral space.

CONTACTS AND LOCATIONS:
Overall Officials: Guanhua Xu, Dr, Principal Investigator — Affiliated 2 Hospital of Nantong University
Locations (1):
- Affiliated 2 Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No